CLINICAL TRIAL: NCT06723834
Title: Psychiatric Service Dogs and Prolonged Exposure Therapy for Military-Connected PTSD: A Randomized Clinical Trial
Brief Title: Service Dogs and Prolonged Exposure Therapy for Military-Connected PTSD
Acronym: SERVES+
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT9425-24-1-0178; CDMRP-PR230987 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Stress Disorders, Post-Traumatic; PTSD; Animal-Human Bonding; Combat Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Human-Animal Bond; Combat Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: (Secondary outcome) PTSD Severity and symptoms via blinded clinician rating, employing the Clinician-Administered PTSD Assessment for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition DSM-V (CAPS-5-R, Range 0-80, Lower scores indicate a better outcome)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD Service Dog + Prolonged Exposure Therapy (Experimental): Participants will receive 12 weeks of Prolonged Exposure once per week with the addition of a service dog
  Interventions: Other: Psychiatric Service Dog; Behavioral: Prolonged Exposure Therapy
- Prolonged Exposure Therapy Alone (Active Comparator): Participants will receive 12 weeks of Prolonged Exposure once per week
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Other: Psychiatric Service Dog — Partnership with a trained service dog for PTSD.
  Arms: PTSD Service Dog + Prolonged Exposure Therapy
Behavioral: Prolonged Exposure Therapy — 12 weeks of Prolonged Exposure once per week.

SUMMARY:
This study investigates the impact of Service Dog partnership on the effectiveness of Prolonged Exposure Therapy. We will learn whether Service Dog partnership in combination with Prolonged Exposure Therapy treatment can help Veterans with PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is common among military Service Members and Veterans (hereafter, "Veterans"). Symptoms of flashbacks, nightmares, and panic attacks can have devastating impacts on Veterans and their families. Suicide and suicidality are also closely linked to PTSD, and the rate of death by suicide among Veterans is nearly double that of the civilian population. PTSD is also difficult to treat. Many Veterans either do not seek treatment at all, or if they start treatment, do not finish. Even if treatment is completed, many Veterans still suffer symptoms and even retain their PTSD diagnosis. There is a critical need to find ways to reduce dropout rates, thus improving the effectiveness of existing, gold-standard treatments and promoting positive outcomes for Veterans and their families.

In their search for effective treatments, some Veterans are turning to add-on interventions for PTSD, such as partnership with a Service Dog. Under the Americans with Disabilities Act (ADA), service dogs are defined as dogs trained to perform specific tasks to mitigate a disability. Service dogs for PTSD are trained in tasks including detecting and alerting to signs of distress to interrupt anxiety and panic attacks and retrieving medication. In addition to trained tasks, service dogs live with the Veterans to provide emotional value as a source of comfort and companionship. Under the ADA guidance, Veterans with PTSD have the legal right to be accompanied by their service dog in public places such as grocery stores, workplaces, and schools. In this study, service dogs will be sourced from participating service dog organizations.

Service Dogs for Veterans are not only increasingly in demand, but a growing body of evidence demonstrates that Service Dogs can significantly improve the lives of Veterans with PTSD. Unfortunately, there is currently no research exploring whether adding a Service Dog will impact the effectiveness of evidence-based PTSD treatments, such as Prolonged Exposure Therapy (PE). Prolonged Exposure Therapy is a gold-standard, frontline treatment for PTSD that is highly effective, but has high rates of dropout.

PE teaches individuals with PTSD to gradually approach trauma-related memories, feelings, and situations that they have been avoiding since their trauma. By confronting these challenges, participants can decrease their PTSD symptoms. PE treatment typically last 12 weeks for 75-90 minutes, once per week.

Initial findings suggest that Service Dogs may help Veterans stay in Prolonged Exposure Therapy resulting in better treatment outcomes. However, some mental health professionals worry that Service Dogs may in fact interfere with treatment goals. This novel study is designed to help understand the impact of Service Dog partnership on the effectiveness of Prolonged Exposure Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Applied for and approved to receive a psychiatric service dog from a service dog organization participating in the study
* Diagnosis of PTSD on the CAPS-5-R

Exclusion Criteria:

* Current service dog
* Current participation in Prolonged Exposure Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptom Severity (Self-report) | 3 months after start of PE
  PTSD Checklist for DSM-5 (PCL-5) Total Score; range 0-80; higher scores indicate worse outcome.

SECONDARY OUTCOMES:
PTSD Symptom Severity (Clinician-assessed) | 3 months after start of PE
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score; range 0-80; higher scores indicate worse outcome.
PTSD Diagnosis | 3 months after start of PE
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Diagnosis; binary
Depression | 3 months after start of PE
  Patient Health Questionnaire (PHQ-9); range 0-27; higher scores indicate worse outcome.
Anxiety | 3 months after start of PE
  Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form 8a; T-score range 37 to 83; 50 indicates the population mean with a standard deviation of 10; minimally important difference greater than or equal to 3 points; higher scores indicate worse outcome.
Emotional affect | 3 months after start of PE
  Bradburn Scale of Psychological Wellbeing (BSPW); range -5 to 5; higher scores indicate better outcome.
Satisfaction with life | 3 months after start of PE
  Satisfaction with Life Scale (SWLS); range 3-35; higher scores indicate better outcome.
Mental health | 3 months after start of PE
  Veterans RAND 12-Item Health Survey Mental Component Score (VR-12 MCS); range 0-100; higher scores indicate better outcome.

OTHER OUTCOMES:
Suicide ideation | 3 months after start of PE
  Beck Scale for Suicide Ideation (BSS) Optimized 6-item Scale; range 0-12; higher score indicates worse outcome.
Suicide cognition | 3 months after start of PE
  Brief Suicide Cognition Scale (B-SCS); range 6-30; higher score indicates worse outcome.
Intrusion (Clinician-assessed) | 3 months after start of PE
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Criterion B Subscale; range 0-20; higher score indicates worse outcome.
Avoidance (Clinician-assessed) | 3 months after start of PE
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Criterion C Subscale; range 0-8; higher score indicates worse outcome.
Cognition and mood (Clinician-assessed) | 3 months after start of PE
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Criterion D Subscale; range 0-28; higher score indicates worse outcome.
Arousal and reactivity (Clinician-assessed) | 3 months after start of PE
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Criterion E Subscale; range 0-24; higher score indicates worse outcome.
Intrusion (Self-report) | 3 months after start of PE
  PTSD Checklist for DSM-5 (PCL-5) Criterion B Subscale; range 0-20; higher score indicates worse outcome.
Avoidance (Self-report) | 3 months after start of PE
  PTSD Checklist for DSM-5 (PCL-5) Criterion C Subscale; range 0-8; higher score indicates worse outcome.
Cognition and mood (Self-report) | 3 months after start of PE
  PTSD Checklist for DSM-5 (PCL-5) Criterion D Subscale; range 0-28; higher score indicates worse outcome.
Arousal and reactivity (Self-report) | 3 months after start of PE
  PTSD Checklist for DSM-5 (PCL-5) Criterion E Subscale; range 0-24; higher score indicates worse outcome.
PE Initiation | 3 months after start of PE
  Binary; whether or not the participant initiated prolonged exposure therapy
PE Session Completion | 3 months after start of PE
  # of prolonged exposure therapy sessions completed (out of 12)
PE Treatment Completion | 3 months after start of PE
  Binary; whether or not the participant completed prolonged exposure therapy
PE Compliance | 3 months after start of PE
  # of inter-session homework assignments completed as part of prolonged exposure therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No